CLINICAL TRIAL: NCT06782009
Title: Metabolic Impact on the Mitochondria-gut Microbiota Axis of Failure to Follow Restrictive Dietary Interventions in Subjects Living With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Laura Alejandra Velázquez Villegas, Investigadora en Ciencias Medicas, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4952
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: dietary restrictions; intermittent fasting; mitochondrial function; gut microbiota; ketogenic diet
MeSH Terms: conditions — Obesity; Intermittent Fasting | interventions — Caloric Restriction; Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: The groups will receive the treatment simultaneously
Who Masked: Investigator
Masking Description: Double single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Calorie Restriction (Experimental): Participants will be provided with a food menu guide for fifteen days with a 30% energy restriction (kcal) according to their usual diet, with a macronutrient distribution of 20-30% protein, 50-60% carbohydrates and 20-30% fat.
  Interventions: Other: Calorie restriction
- Intermittent fasting 16/8 (Experimental): Participants will be provided with a food menu guide for fifteen days with an energy intake according to the energy expenditure determined by indirect calorimetry with normal distribution of macronutrients. Intermittent fasting will be used with a time-restricted model of 16:8. For 16 hours, they will not be able to eat or drink calories. In the other 8 hours, they need to adhere to the energy-restricted diet.
  Interventions: Other: Intermittent fasting 16/8
- Ketogenic diet (Experimental): Participants will be provided with a food menu guide for 15 days with an energy intake according to the energy expenditure determined by indirect calorimetry, with the following distribution of macronutrients: 20-25% protein, 5-10% carbohydrates, 70-80% fat.
  Interventions: Other: Ketogenic diet

INTERVENTIONS:
Other: Calorie restriction — Participants will be provided with a food menu guide for fifteen days with a 30% energy restriction (kcal) according to their usual diet, with a macronutrient distribution of 20-30% protein, 50-60% carbohydrates and 20-30% fat.
  Arms: Calorie Restriction
Other: Intermittent fasting 16/8 — Participants will be provided with a food menu guide for fifteen days with an energy intake according to the energy expenditure determined by indirect calorimetry with normal distribution of macronutrients. Intermittent fasting will be used with a time-restricted model of 16:8. For 16 hours, they will not be able to eat or drink calories. In the other 8 hours, they need to adhere to the energy-restricted diet.
  Arms: Intermittent fasting 16/8
Other: Ketogenic diet — Participants will be provided with a food menu guide for 15 days with an energy intake according to the energy expenditure determined by indirect calorimetry, with the following distribution of macronutrients: 20-25% protein, 5-10% carbohydrates, 70-80% fat.
  Arms: Ketogenic diet

SUMMARY:
Nutritional interventions with dietary restrictions have become highly popular for promoting weight and body fat loss; In addition, they are largely associated with the improvement and preservation of mitochondrial function as well as the changes they generate in the composition of the gut microbiota and microbial metabolites. During obesity, mitochondrial dysfunction in monocytes can increase low-grade inflammation and contribute to alterations in various metabolic tissues. There have been many studies that have been dedicated to describing the benefits and mechanisms of the use of restrictive interventions, but few have focused on further monitoring and evaluating the metabolic changes that occur due to the lack of follow-up of the use of these interventions, where subjects resume eating patterns with energy overload. behavior that happens in the vast majority of patients, so keeping mitochondria in good condition is a key aspect of maintaining health. The present project aims to study the metabolic changes that are generated by the lack of follow-up of restrictive dietary interventions, focusing on the effects produced in mitochondrial function evaluated in monocytes isolated from peripheral blood and the impact that the composition of the intestinal microbiota is generated from the metabolites produced, affecting as a consequence the inflammatory state of the host. A randomized controlled clinical trial will be carried out where the selected participants will be assigned by lottery to one of the 3 nutritional interventions for 8 weeks, then the participants will be followed up at 8, 16 and 24 weeks after the intervention has ended. Anthropometric and biochemical parameters, resting energy expenditure, blood pressure, oxidative stress markers, metabolomics, gut microbiota composition, and mitochondrial function will be evaluated during follow-up.

DETAILED DESCRIPTION:
The study consists of an open-label randomized controlled clinical trial. The selected subjects will be men or women over 18 years of age with a body mass index (BMI) greater than or equal to 30 kg/m2, who meet the selection criteria, the subjects who will be randomly assigned to one of 3 dietary intervention groups. The study consisted of a dietary intervention with a duration of 8 weeks and a follow-up of 24 weeks after dietary intervention.

The intervention groups will be as follows:

1. Calorie-restricted diet: Dietary recommendations will be given restricting 30% in energy (kcal) according to their usual diet with normal macronutrient distribution (20-30% protein, 50-60% carbohydrates, 20-30% fats).
2. Intermittent fasting diet: Dietary recommendations will be given according to the energy expenditure determined by indirect calorimetry with normal macronutrient distribution. Intermittent fasting will be used with a time-restricted model of 16:8. For 16 hours, they will not be able to eat or drink calories. In the other 8 hours, they need to adhere to the energy-restricted diet.
3. Ketogenic diet: Recommendation will be given according to the energy expenditure determined by indirect calorimetry, with the following distribution of macronutrients: 20-25% protein, 5-10% carbohydrates, 70-80% fat.

Participants with calorie-restriction, intermittent fasting, or ketogenic diet dietary intervention will be provided with a food menu guide for fifteen days. After 8 weeks of the assigned intervention, patients will be provided with general dietary recommendations and will be invited to three more follow-up visits at 8, 16 and 24 weeks post-intervention. In addition, all participants will be provided with general recommendations for a physical activity plan for people living with obesity.

To evaluate adherence to treatment, participants will be asked to fill out 2 logbooks every two weeks (1 during the week and 1 for the weekend) in which they must record the type, amount and place where they consumed the food at each feeding time. They will also be called once a week for a 24-hour reminder. Participants on the ketogenic diet will be given test strips to measure ketones in urine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female.
* Adults >18 years of age.
* BMI ≥ 30 kg/m2

Exclusion Criteria:

* Patients with any type of diabetes.
* Patients with high blood pressure.
* Patients with acquired diseases secondarily producing obesity and diabetes.
* Patients who have suffered a cardiovascular event.
* Patients who at the screening visit presented glucose values greater than 126 mg/dL, triglycerides greater than 350 mg/dL, cholesterol greater than 300mg/dL and/or creatinine greater than 1.2 mg/dL in men and greater than 1 mg/dL in women.
* Patients with gastrointestinal diseases.
* Weight loss > 3 kg in the last 3 months.
* Catabolic diseases such as cancer and acquired immunodeficiency syndrome.
* Pregnancy status.
* Positive smoking.
* History of major surgery requiring general or regional anesthesia, respiratory support, and involving a recovery time longer than 2 weeks, such as surgeries of the abdomen (bowel resection), chest, head, and neck.
* Diagnosis of Anxiety and Depression as Determined by the HADS Scale
* Drug treatment:
* Antihypertensive drugs or treatment
* Treatment with hypoglycemic agents or insulin and antidiabetic drugs.
* Treatment with statins, fibrates or other drugs to control dyslipidemia.
* Use of antibiotics in the three months prior to the study.
* Use of steroid drugs, chemotherapy, immunosuppressants, or radiation therapy.
* Anorexigenic or that accelerate weight loss such as sibutramine or orlistat.
* Supplements with any of the functional foods used in the study.
* Probiotic, prebiotic or symbiotic supplements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial function | baseline to 8, 16, 24 and 32 weeks
  Change in mitochondrial function determined by measuring the oxygen consumption rate (OCR) in isolated monocytes

SECONDARY OUTCOMES:
Gut microbiota composition | baseline to 8, 16 and 32 weeks
  Change in gut microbiota composition determined by bacterial abundance obtained after taxonomy assignment.
Body weight measurement | baseline to 8, 16, 24 and 32 weeks
  Change in body weight determined by scale.
Glucose concentration | baseline to 8, 16, 24 and 32 weeks
  Change in glucose in the serum determined by autoanalyzer.
Cholesterol concentration | baseline to 8, 16, 24 and 32 weeks
  Change in cholesterol in the serum determined by autoanalyzer.
HDL cholesterol concentration | baseline to 8, 16, 24 and 32 weeks
  Change in HDL cholesterol in the serum determined by autoanalyzer.
LDL cholesterol concentration | baseline to 8, 16, 24 and 32 weeks
  Change in LDL cholesterol in the serum determined by autoanalyzer.
Triglycerides concentration | baseline to 8, 16, 24 and 32 weeks
  Change in triglycerides in the serum determined by autoanalyzer.
Insulin concentration | baseline to 8, 16, 24 and 32 weeks
  Change in insulin in the serum determined by ELISA kit.
Leptin concentration | baseline to 8, 16, 24 and 32 weeks
  Change in leptin in the serum determined by ELISA kit.
Interleukins concentration | baseline to 8, 16, 24 and 32 weeks
  Change in interleukins in the serum determined by ELISA kit.
C-reactive protein concentration | baseline to 8, 16, 24 and 32 weeks
  Change in C-reactive protein in the serum determined by autoanalyzer.
TNF-a concentration | baseline to 8, 16, 24 and 32 weeks
  Change in TNF-a in the serum determined by ELISA kit.
Alpha diversity of gut microbiota | baseline to 8, 16 and 32 weeks
  Shanon index to indicate alpha diversity of gut microbiota from the feces
Beta diversity of gut microbiota | baseline to 8, 16 and 32 weeks
  Principal component analysis to indicate alpha diversity of gut microbiota from the feces
Fat mass percentage | baseline to 8, 16, 24 and 32 weeks
  Fat mass percentage determined by multifrequency electrical bioimpedance.
Lean mass percentage | baseline to 8, 16, 24 and 32 weeks
  Lean mass percentage determined by multifrequency electrical bioimpedance.
Skeletal muscle mass percentage | baseline to 8, 16, 24 and 32 weeks
  Skeletal muscle mass percentage determined by multifrequency electrical bioimpedance.
Change of metabolites in serum | baseline to 8, 16 and 32 weeks
  Change of metabolites in serum determined by un-targeted metabolomics using Liquid chromatography/ Mass spectrometry analysis (LC/MS).
Change of metabolites in feces | baseline to 8, 16 and 32 weeks
  Change of metabolites in feces determined by un-targeted metabolomics using Liquid chromatography/ Mass spectrometry analysis (LC/MS).
Determination of valvular function | baseline to 8 weeks
  Doppler venous ultrasound will be performed with the MX7 equipment of the Shenzhen Mindray Bio-Medical Electronics Co., LTD to determine the valvular function of the great saphenous vein, small saphenous vein, junction femoral saphenous vein, femoral vein, popliteal vein, measuring their dimensions and the level of venous reflux.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Velazquez Villegas, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (2):
- Mexico (2):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Tlalpan
  - Departamento de Fisiología de la Nutrición. Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City

IPD SHARING:
Plan to Share IPD: No
Data may be shared after publication.

REFERENCES:
- [Background] Guevara-Cruz M, Hernandez-Gomez KG, Condado-Huerta C, Gonzalez-Salazar LE, Pena-Flores AK, Pichardo-Ontiveros E, Serralde-Zuniga AE, Sanchez-Tapia M, Maya O, Medina-Vera I, Noriega LG, Lopez-Barradas A, Rodriguez-Lima O, Mata I, Olin-Sandoval V, Torres N, Tovar AR, Velazquez-Villegas LA. Intermittent fasting, calorie restriction, and a ketogenic diet improve mitochondrial function by reducing lipopolysaccharide signaling in monocytes during obesity: A randomized clinical trial. Clin Nutr. 2024 Aug;43(8):1914-1928. doi: 10.1016/j.clnu.2024.06.036. Epub 2024 Jul 5. PMID 39003957
- [Background] Guevara-Cruz M, Hernandez-Gomez KG, Condado-Huerta C, Gonzalez-Salazar LE, Pena-Flores AK, Pichardo-Ontiveros E, Serralde-Zuniga AE, Sanchez-Tapia M, Maya O, Medina-Vera I, Noriega LG, Lopez-Barradas A, Rodriguez-Lima O, Mata I, Olin-Sandoval V, Torres N, Tovar AR, Velazquez-Villegas LA. Reply - Letter to the editor- enhancing understanding of dietary interventions in obesity: Insights and recommendations for future research. Clin Nutr. 2024 Sep;43(9):2211-2213. doi: 10.1016/j.clnu.2024.08.006. Epub 2024 Aug 13. No abstract available. PMID 39173436